CLINICAL TRIAL: NCT04748575
Title: Effect of Acute Acai Berry Supplementation on Post-prandial Glycaemia in Healthy Adults: a Randomised Controlled Study
Brief Title: Effect of Acai Berry Consumption on Blood Glucose Levels in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Mary's University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: SMU_ETHICS_2020-21_111
Record Dates: First submitted 2021-02-04; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Post-prandial Glycaemia
Keywords: Acai (Euterpe oleracea), acute

STUDY DESIGN:
Intervention Model Description: Randomised double-blind crossover
Who Masked: Participant, Investigator
Masking Description: Smoothies were prepared by the Laboratory Technician and blinded from the participant and investigator. Acai and placebo smoothies were matched nutritionally including for carbohydrate, total sugars, protein, fat and fibre. Additionally, the smoothies were matched for colour, taste and temperature and were served in opaque containers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acai smoothie consumption (Experimental): Participants (n=5) in this arm were randomly allocated to consume the acai smoothie at the first intervention. After a 7 day wash-out period, the participants consumed the placebo smoothie.
  Interventions: Dietary Supplement: Acai smoothie
- Placebo smoothie consumption (Experimental): Participants (n=5) in this arm were randomly allocated to consume the placebo smoothie at the first intervention. After a 7 day wash-out period, the participants consumed the acai smoothie.
  Interventions: Dietary Supplement: Placebo smoothie

INTERVENTIONS:
Dietary Supplement: Acai smoothie — Smoothie containing 150g acai pulp
  Arms: Acai smoothie consumption
Dietary Supplement: Placebo smoothie — Control smoothie matched nutritionally (macronutrients) and sensorially to the acai smoothie.
  Arms: Placebo smoothie consumption

SUMMARY:
Type 2 Diabetes Mellitus is a chronic disease that results in hyperglycaemia. This study aimed to identify whether the anthocyanins contained in acai berries can mitigate postprandial glycaemia in healthy adults when consumed in conjunction with carbohydrate. Study design was double blind randomised crossover with glycaemic levels assessed via capillary blood samples taken at baseline and over a 2 hour post-prandial period.

DETAILED DESCRIPTION:
Type 2 Diabetes Mellitus (T2DM) is a group of chronic metabolic disorders, characterised by insulin resistance and relative insulin deficiency, that results in hyperglycaemia. In the UK an estimated 4.3m people live with T2DM, and it is a major cause of kidney failure, heart attacks, stroke, blindness and lower limb amputation. The primary digestive enzymes that affect carbohydrate digestion and hence postprandial glycaemic levels have been identified as α-amylase and α-glucosidase. Inhibition of these enzymes therefore reduces the rate of glucose absorption and is the principle behind T2DM medications such as acarbose, miglitol and voglibose. Whilst acai berries have been found to be rich in α-amylase and α-glucosidase, no research has been conducted on healthy adults to ascertain whether the consumption of acai berries in conjunction with carbohydrate mitigates the rise in postprandial glycaemia.

10 participants were recruited for a double blind randomised crossover study where participants consumed smoothies containing either acai or placebo after 10 hours of fasting. Capillary blood samples were taken at baseline then at 30 minutes intervals until 2 hours after consumption. The study included data for sex (female/male), age (years), weight (kg), height (cm), body mass index (kg/m2) and blood glucose (mmol/l). All data collection, smoothies preparation, smoothies consumption and blood sampling procedures were completed at St Mary's University during the period November-December 2020. Statistical analysis was conducted on the data for postprandial glycaemic response to ascertain whether the consumption of acai mitigated the glycaemic response relative to the placebo.

ELIGIBILITY:
Inclusion Criteria:

• BMI of 18.5 - 24.9 kg/m2.

Exclusion Criteria:

* Known allergy to acai/berries or lactose.
* Pregnant or lactating.
* Alcohol/drug dependency.
* Smoking.
* Currently on an energy-restriction diet or have had a body weight change >10% in last 2 months.
* Eating disorders.
* Diagnosed with diabetes or another chronic condition.
* Taking chronic medication.
* Allergy to any of materials used in, or an unsurmountable fear of, the finger-prick procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Blood glucose | Baseline to 120 minutes after intervention.
  Finger capillary sample collected by micro cuvette (Glucose 201, HemoCue, UK) and analysed electronically (HemoCue 201+, HemoCue,UK).

CONTACTS AND LOCATIONS:
Locations (1):
- St Marys University, London, United Kingdom